CLINICAL TRIAL: NCT05785572
Title: Study on the of Preoperative Analgesia With Radiofrequency of Suprascapular Nerve Versus Intraoperative Interscalene Block on Postoperative Pain in Shoulder Rerverse Arthroplasty Surgery
Brief Title: Effect of Radiofrequency of Suprascapular Nerve in Shoulder Reverse Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAP_PIH_20
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Tear Arthropathy; Post Operative Pain
Keywords: rotator cuff arthropathy; reverse shoulder arthroplasty; supraescapular nerve radiofrecuency; post operative pain
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized clinical trial with two groups of study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency group (Experimental): Patient group that undergoes Radiofrequency of supraescapular nerve before shoulder arthroplasty surgery
  Interventions: Procedure: supraescapular nerve radiofrequency
- Interscalenic braquial plexus block group (Active Comparator): Interscalenic braquial plexus block done at the moment of the surgery.
  Interventions: Procedure: interescalenic braquial plexus

INTERVENTIONS:
Procedure: supraescapular nerve radiofrequency — supraescapular nerve radiofrequency or interescalenic braquial plexus for pain control in shoulder arthroplasty surgery
  Arms: Radiofrequency group
Procedure: interescalenic braquial plexus — supraescapular nerve radiofrequency or interescalenic braquial plexus for pain control in shoulder arthroplasty surgery
  Arms: Interscalenic braquial plexus block group

SUMMARY:
The purpuse of this study is to asses if the pulsed radiofrecuency of the supraescapular nerve and accesory nerve have the same or superior efectivity controlling the acute postoperative pain than interscalenic braquial plexus block

DETAILED DESCRIPTION:
This is a randomized, double-blind trial that compares the effect in postoperative pain of pulsed radiofrecuency of the supraescapular nerve carried out at least two to four weeks before reverse total shoulder arthroplasty surgery with interscalenic braquial plexus block done at the moment of the surgery. All the patients received conventional general anaesthesia and multimodal postoperative analgesia with additional patient-controlled rescue analgesics were prescribed

ELIGIBILITY:
Inclusion criteria:

* Over 18 y.o.
* Cronic pain (more than 3 months) due to rotator cuff arthropathy
* VAS higher than 4
* Decrease Constant score
* Conservative treatment (physiotherapy and NSAIs) unsuccessful

Exclusion criteria:

* psychiatric illness
* drug abuse.
* previous surgeries.
* acute traumatic pathology or ethiology different from rotator cuff arthropathy
* pacemaker
* infectious process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogical scale | periodical measurements of pain, inmediate preoperative pain up to three months postoperative
  Postoperative acute pain measurement. From 0 to 10, Zero means no pain and ten would be the worse pain that the paitient could feel.

SECONDARY OUTCOMES:
Visual analogical scale | 3 months postop. until 1 year postop
  chronic pain after surgery. From 0 to 10, Zero means no pain and ten would be the worse pain that the paitient could feel.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Lopez Millan, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain